CLINICAL TRIAL: NCT01636752
Title: Effectiveness of Internet-based Depression Treatment
Acronym: EVIDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Philipp Klein, Coordinating Investigator, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVIDENT Trial
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Mild to Moderate Depressive Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deprexis (Experimental): Online self-help with and without e-mail-support
  Interventions: Behavioral: Deprexis
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Deprexis — Online self-help with and without e-mail-support
  Arms: Deprexis

SUMMARY:
Care for people suffering from depressive symptoms should be given in a step-wise approach. One first step can be the provision of self-help material. Online self-help is an innovative way of providing self-help. The investigators want to study the effect of an interactive online self-help-program (Deprexis) in the treatment of mild to moderate depressive symptoms. Participants will be randomised to either twelve weeks of online-self help or a waiting-list control. Symptoms of depression and other aspects will be assessed over a one year period. Thereafter the controls will also receive online-self help. The investigators hypothesise that online self-help is superior to the control condition in alleviating depressive symptoms and preventing full blown depression.

DETAILED DESCRIPTION:
This study is supported by the German Ministry of Health (BMG) and is a collaborative project of Universität Bern (PD Dr. Thomas Berger), Charité Berlin (PD Dr. Matthias Rose), Universität Bielefeld (Prof. Dr. Wolfgang Greiner), Universität Hamburg (Prof. Dr. Steffen Moritz, Prof. Dr. Bernd Löwe), GAIA AG Hamburg (Dr. Björn Meyer), Universität Tübingen (Prof. Dr. Martin Hautzinger) and Universität Trier (Prof. Dr. Wolfgang Lutz).

ELIGIBILITY:
Inclusion Criteria:

* PHQ>4 and <15

Exclusion Criteria:

* acute suicidality
* psychotic d/o, bipolar d/o or other severe psychiatric d/o

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Personal Health Questionnaire (PHQ-9) | 12 wks

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression (HRSD) | 12 wks, 6 mths, 12 mths
Quick Inventory of Depressive Symptoms (QIDS) | 12 wks, 6 mths, 12 mths
Personal Health Questionnaire (PHQ-9) | 6 mths, 12 mths

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Charité Berlin, Berlin
  - Universität Bielefeld, Bielefeld
  - Universität Hamburg, Hamburg
  - Universität Lübeck, Lübeck

REFERENCES:
- [Background] Klein JP, Berger T, Schroder J, Spath C, Meyer B, Caspar F, Lutz W, Greiner W, Hautzinger M, Rose M, Grafe V, Hohagen F, Andersson G, Vettorazzi E, Moritz S. The EVIDENT-trial: protocol and rationale of a multicenter randomized controlled trial testing the effectiveness of an online-based psychological intervention. BMC Psychiatry. 2013 Sep 28;13:239. doi: 10.1186/1471-244X-13-239. PMID 24074299
- [Result] Klein JP, Berger T, Schroder J, Spath C, Meyer B, Caspar F, Lutz W, Arndt A, Greiner W, Grafe V, Hautzinger M, Fuhr K, Rose M, Nolte S, Lowe B, Anderssoni G, Vettorazzi E, Moritz S, Hohagen F. Effects of a Psychological Internet Intervention in the Treatment of Mild to Moderate Depressive Symptoms: Results of the EVIDENT Study, a Randomized Controlled Trial. Psychother Psychosom. 2016;85(4):218-28. doi: 10.1159/000445355. Epub 2016 May 27. PMID 27230863
- [Derived] Nolte S, Busija L, Berger T, Meyer B, Moritz S, Rose M, Schroder J, Spath-Nellissen C, Klein JP. Do sociodemographic variables moderate effects of an internet intervention for mild to moderate depressive symptoms? An exploratory analysis of a randomised controlled trial (EVIDENT) including 1013 participants. BMJ Open. 2021 Jan 26;11(1):e041389. doi: 10.1136/bmjopen-2020-041389. PMID 33500282
- [Derived] Probst T, Berger T, Meyer B, Spath C, Schroder J, Hohagen F, Moritz S, Klein JP. Social phobia moderates the outcome in the EVIDENT study: A randomized controlled trial on an Internet-based psychological intervention for mild to moderate depressive symptoms. J Consult Clin Psychol. 2020 Jan;88(1):82-89. doi: 10.1037/ccp0000441. Epub 2019 Nov 4. PMID 31682137
- [Derived] Arndt A, Lutz W, Rubel J, Berger T, Meyer B, Schroder J, Spath C, Hautzinger M, Fuhr K, Rose M, Hohagen F, Klein JP, Moritz S. Identifying change-dropout patterns during an Internet-based intervention for depression by applying the Muthen-Roy model. Cogn Behav Ther. 2020 Jan;49(1):22-40. doi: 10.1080/16506073.2018.1556331. Epub 2019 Feb 5. PMID 30721109
- [Derived] Schroder J, Berger T, Meyer B, Lutz W, Spath C, Michel P, Rose M, Hautzinger M, Hohagen F, Klein JP, Moritz S. Impact and change of attitudes toward Internet interventions within a randomized controlled trial on individuals with depression symptoms. Depress Anxiety. 2018 May;35(5):421-430. doi: 10.1002/da.22727. Epub 2018 Feb 28. PMID 29489038
- [Derived] Klein JP, Spath C, Schroder J, Meyer B, Greiner W, Hautzinger M, Lutz W, Rose M, Vettorazzi E, Andersson G, Hohagen F, Moritz S, Berger T. Time to remission from mild to moderate depressive symptoms: One year results from the EVIDENT-study, an RCT of an internet intervention for depression. Behav Res Ther. 2017 Oct;97:154-162. doi: 10.1016/j.brat.2017.07.013. Epub 2017 Jul 21. PMID 28797829
- [Derived] Klein JP, Gamon C, Spath C, Berger T, Meyer B, Hohagen F, Hautzinger M, Lutz W, Vettorazzi E, Moritz S, Schroder J. Does recruitment source moderate treatment effectiveness? A subgroup analysis from the EVIDENT study, a randomised controlled trial of an internet intervention for depressive symptoms. BMJ Open. 2017 Jul 13;7(7):e015391. doi: 10.1136/bmjopen-2016-015391. PMID 28710212